CLINICAL TRIAL: NCT01475487
Title: A Comparison of Ultrasound Versus Digital Palpation Guided Cricothyrotomy in Subjects With Poorly Defined Anatomical Landmarks
Brief Title: Ultrasound Guided Versus Palpation Guided Cricothyrotomy With Poorly Defined Anatomical Landmarks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Principal Investigator, Dr. Naveed Siddiqui, Assistant Professor, Samuel Lunenfeld Research Institute, Mount Sinai Hospital
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: CUS-2010
Record Dates: First submitted 2011-11-03; First posted 2011-11-21 (Estimated); Results first posted 2015-06-25 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-06

CONDITIONS: Airway Management

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cricothyrotomy using Digital Palpation (Active Comparator): Group-1 will perform Cricothyrotomy using conventional digital palpation technique
  Interventions: Procedure: Utrasound guided cricothyrotomy
- Ultrasound guided cricothyrotomy group (Experimental): Group-2 Ultrasound guided cricothyrotomy
  Interventions: Procedure: Utrasound guided cricothyrotomy

INTERVENTIONS:
Procedure: Utrasound guided cricothyrotomy — Utrasound guided cricothyrotomy

SUMMARY:
Inability to provide oxygen to the patient remains the most fearful anesthesia-related mishap. Cricothyrotomy (CT) is an infrequently performed but life saving procedure for an anesthesiologist, who is encountered with this situation. The current method of cricothyrotomy relies on digital palpation (DP). Several patient populations, including morbidly obese, short neck, radiation to and previous neck surgeries, have difficult landmarks for this procedure. Ultrasound (US) technology has been used in the past to visualize landmarks for cricothyrotomy, but there is no study which has examined the role of ultrasound in patients who have obscure landmarks. There is no data related to the performance of ultrasound guided cricothyrotomy in these patients. In this study, we aimed to determine the outcomes of CT performed on human cadavers using US-guidance, compared to conventional DP, of anatomical landmarks. In particularly, complication rates, failure to cannulate, correct placement of the device and insertion time of CT were assessed.

DETAILED DESCRIPTION:
For each cadaver - epidemiological data (age, sex) and morphometric data (Body Mass Index, neck circumference, thyromental distance)

The primary outcome measure was the complication rate as assessed by the severity of injuries; defined as the incidence and severity of posterior laryngeal and tracheal wall injuries, as graded by two anesthesiologists using the grading system described by Murphy et al,( none (no injury); mild (< 5 mm laceration); moderate (> 5mm laceration or partial puncture); severe (> 10 mm laceration or full puncture)). For clinical relevance and analysis of data we dichotomized the scale to none-mild and moderate - severe injuries.

The secondary outcomes include: 1) insertion time, measured in seconds (s) from the time of palpation of the skin to insertion of the Portex device in the trachea; 2) failure, with a 'failure' defined as any attempt in which the trachea was not cannulated, or which required > 300 s to perform; and 3) correct land-marking, defined as having the Portex device inserted via the CM.

ELIGIBILITY:
Inclusion Criteria:

* Residents who are novice to the application of ultrasound in difficult airway scenarios
* Cadavers with difficult and imposible landmarks identification

Exclusion Criteria:

* Anethesiologist with previous experience in CT, manual or ultrasound assisted
* Patients with easily identifiable landmarks

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2011-04; Primary Completion 2011-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naveed Siddiqui, MD, Principal Investigator — Mount Sinai Hospital Department of Anesthesia and Pain Management

RESULTS

PARTICIPANT FLOW:
Groups:
- Cricothyrotomy Using Digital Palpation: Group-1 will perform cricothyrotomy using conventional digital palpation technique
  The identification of the cricothyroid membrane by digital palpation was performed by using the index and third fingers of the non-dominant hand. The thyroid cartilage was first palpated in the midline starting from cephalad and moving caudally until the cricoid cartilage is palpated. The is the space between the inferior border of the thyroid cartilage and the superior border of the cricoid cartilage
- Ultrasound Guided Cricothyrotomy Group: Group-2 Ultrasound guided cricothyrotomy A 15-10 mHz linear probe (MicroMaxx system, Sonosite Canada Inc, Markham, Ontario, Canada) was used to obtain sonographic images of anatomical landmarks on cadaveric necks as described by Kristensen.
  The participants held the linear high-frequency transducer in their non-dominant hand and placed themselves on the right side of the cadaver facing towards the head of the cadaver. Then they placed the US probe transversely over the cadaver's neck just above the suprasternal notch in order to visualize the trachea. The transducer was then moved laterally to the patient's right side until the right border of the transducer was superficial to the midline of the trachea. During this movement it was ensured that the right end of the transducer was kept in the midline of the trachea while the left end of the transducer was rotated into the sagittal plane resulting in a longitudinal scan of the midline of the trachea.
Period: Overall Study
Arm/Group | Cricothyrotomy Using Digital Palpation | Ultrasound Guided Cricothyrotomy Group
Started | 25 | 25
Completed | 23 | 24
Not Completed | 2 | 1
Not completed — had to leave early for personal reasons | 2 | 1

BASELINE CHARACTERISTICS:
Population: Characteristics of participants and human cadavers
Groups:
- Total: Total of all reporting groups
Arm/Group | Cricothyrotomy Using Digital Palpation | Ultrasound Guided Cricothyrotomy Group | Total
Number analyzed (Participants) | 23 | 24 | 47
Age, Customized [Number] | NA — Age was not collected for this study | NA — Age was not collected for this study | NA — Total not calculated because data are not available (NA) in one or more arms.
Sex: Female, Male [Count of Participants; unit: Participants] — Gender description is for Cadvaers only
  Participants
    Female | 11 | 17 | 28
    Male | 12 | 7 | 19
Neck circumference [Mean (Standard Deviation); unit: Centimeters] | 21.35 (1.92) | 21.54 (1.74) | 21.45 (1.74)
Landmark grade [Number; unit: participants] — Landmark grade indicate the difficulty in identification of anatomical landmarks on the cadavers. Higher grades indicate a greater difficulty in identification
  participants
    Grade-2 | 11 | 9 | 20
    Grade-3 | 8 | 8 | 16
    Grade-4 | 4 | 7 | 11
Years post graduate trainee level [Number; unit: Participants]
  POST GRADUATE YEAR-1 | 4 | 7 | 11
  POST GRADUATE YEAR-2 | 7 | 4 | 11
  POST GRADUATE YEAR-3 | 4 | 2 | 6
  POST GRADUATE YEAR-4 | 2 | 3 | 5
  POST GRADUATE YEAR-5 | 2 | 4 | 6
  FELLOWS | 4 | 4 | 8

OUTCOME MEASURES:

1. Secondary Outcome: Insertion Time
Description: Defined as palpation of the skin to completion of procedure- cannula in trachea.
Time Frame: less than 5 minutes from starting of procedure
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Cricothyrotomy Using Digital Palpation | Ultrasound Guided Cricothyrotomy Group
Number analyzed (Participants) | 23 | 24
seconds | 110.48 (46.94) | 196.13 (60.64)
Statistical Analysis 1: Comparison: Cricothyrotomy Using Digital Palpation vs Ultrasound Guided Cricothyrotomy Group; Test type: Non-Inferiority or Equivalence — A sample size of 21 participants per group was required to detect a 40% absolute difference in the complication rate between DP and US guided techniques assuming a 45% complication rate in the DP (control) group and using the Fisher's exact test for the comparison of independent proportions. A total of 23 and 24 participants were recruited in the DP and US group, respectively; p < 0.01, Fisher Exact

2. Primary Outcome: The Primary Outcome Measure Was the Complication Rate Asssed as the Number of Participants Causing Injuries
Description: The primary outcome measure was the complication rate as assessed by the severity of injuries; defined as the incidence and severity of posterior laryngeal and tracheal wall injuries, as graded by two anesthesiologists using the grading system described by Murphy et al,( none (no injury); mild (< 5 mm laceration); moderate (> 5mm laceration or partial puncture); severe (> 10 mm laceration or full puncture)).
Time Frame: On avergae less than 300 seconds
Measure: Number; unit: Participants
Arm/Group | Cricothyrotomy Using Digital Palpation | Ultrasound Guided Cricothyrotomy Group
Number analyzed (Participants) | 23 | 24
Participants
  None - Mild Grade-1-4(n=23,24) | 6 | 18
  Moderate-severe Grade 1-4(n=23,24) | 17 | 6
  None -Mild Grade 3-4(n=12,15) | 0 | 10
  Moderate-severe Grade 3-4(n=12,15) | 12 | 5
Statistical Analysis 1: Comparison: Cricothyrotomy Using Digital Palpation vs Ultrasound Guided Cricothyrotomy Group; Test type: Superiority or Other; p = 0.001, Fisher Exact; Risk Ratio (RR) = 2.88, 95% CI 2-sided [1.39 to 5.94] — Risk of injury ( none-mild vs moderate -severe) for all participants
Statistical Analysis 2: Comparison: Cricothyrotomy Using Digital Palpation vs Ultrasound Guided Cricothyrotomy Group; Grade 3-4 comparison of None-mild and moderate-severe; Test type: Superiority or Other; p < 0.001, Fisher Exact

3. Secondary Outcome: Number of Attempts
Description: Number of attempts were defined as an actual attempt to cannulate trachea or layrnx of the cadavers by the participants.
Time Frame: not more than 300 seconds
Measure: Number; unit: participants
Arm/Group | Cricothyrotomy Using Digital Palpation | Ultrasound Guided Cricothyrotomy Group
Number analyzed (Participants) | 23 | 24
participants
  attempt 1 | 20 | 19
  attempt 2 | 3 | 5
Statistical Analysis 1: Comparison: Cricothyrotomy Using Digital Palpation vs Ultrasound Guided Cricothyrotomy Group; Test type: Superiority or Other; p = 0.701, Fisher Exact; Risk Ratio (RR) = 0.91, 95% CI 2-sided [0.12 to 2.72] — This is the risk ratio for 1 vs 2 attempts

4. Secondary Outcome: Correct Landmarking
Description: Correct landmarking by all participants between the ultrasound and digital palpation group
Time Frame: less than 300 seconds
Measure: Number; unit: participants
Arm/Group | Cricothyrotomy Using Digital Palpation | Ultrasound Guided Cricothyrotomy Group
Number analyzed (Participants) | 23 | 24
participants
  yes (grade1-4) | 9 | 15
  no (grade 1-4) | 14 | 9
  Yes ( Grade3-4) | 1 | 7
  No ( Grade3-4) | 11 | 8
Statistical Analysis 1: Comparison: Cricothyrotomy Using Digital Palpation vs Ultrasound Guided Cricothyrotomy Group; Comparison for Grade 3-4; Test type: Superiority or Other; p = 0.043, Fisher Exact; Risk Ratio (RR) = 5.60, 95% CI 2-sided [0.79 to 39.48]

ADVERSE EVENTS:
Description: Serious and other non serious adverse events were not collected
Arm/Group | Cricothyrotomy Using Digital Palpation | Ultrasound Guided Cricothyrotomy Group
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes